CLINICAL TRIAL: NCT07209527
Title: Evaluation of Truway Health-Sourced Portable Diagnostic Devices for Early Detection of Chronic Conditions in Outpatient Primary Care Settings: A Prospective Interventional Study
Brief Title: Truway Diagnostic Tools in Primary Care
Acronym: TruDxPC
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Truway Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: TRHW-DX-001
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Chronic Disease; Type 2 Diabetes Mellitus (T2DM), Obesity, Overweight; Hypertension; Cardiovascular Disease Acute; Hyperlipidemia; Chronic Kidney Disease (CKD), Stages 3-4 Exercise Tolerance / Functional Capacity Vascular Health / Arterial Stiffness Fatigue in CKD; Peripheral Artery Disease; Metabolic Syndrome; Prediabetes
Keywords: Portable Diagnostic Devices; Ultrasound; Blood Glucose Monitoring; Chronic Disease Management; Early Detection; Primary Care; Interventional Study; Truway Health; Diabetes; Cardiovascular Disease; Hypertension; Obesity; Metabolic Syndrome; Outpatient Care; Clinical Trial
MeSH Terms: conditions — Chronic Disease; Diabetes Mellitus, Type 2; Obesity; Overweight; Hypertension; Hyperlipidemias; Renal Insufficiency, Chronic; Peripheral Arterial Disease; Metabolic Syndrome; Prediabetic State; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This study employs an Interventional Study Model designed as a parallel assignment with a sequential enrollment approach. Participants (n=200) will be randomly assigned to one of two groups: an intervention group utilizing Truway Health-sourced portable diagnostic devices (ultrasound and blood glucose monitors) under supervised primary care protocols, or a control group receiving standard care without these tools. The parallel assignment ensures simultaneous comparison of outcomes between the groups over the 6-month intervention period.The sequential enrollment strategy involves staged recruitment, beginning with 100 participants at the initial site (Truway Health Clinical Research Center, New York, NY) starting February 1, 2026, followed by an additional 100 participants at a planned Miami, FL site pending successful interim analysis (targeted for May 2026). This phased approach allows for monitoring of device performance and safety data before expanding, with adjustments to protocols
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: Yes

ARMS (2):
- Intervention Group with Truway Diagnostic Devices (Experimental): Participants (n=100) will use Truway Health-sourced portable ultrasound and blood glucose monitors under supervised primary care protocols. The intervention aims to enhance early detection of chronic conditions (e.g., diabetes, cardiovascular disease) over 6 months, with follow-ups at 3 and 6 months to assess diagnostic accuracy and clinical outcomes. Devices are calibrated and provided by Truway Health, Inc., with training for care providers.
  Interventions: Device: Truway Portable Ultrasound Device; Device: Truway Blood Glucose Monitor; Drug: Standard Oral Hypoglycemic Agent
- Control Group with Standard Care (Active Comparator): Participants (n=100) will receive standard care without Truway diagnostic devices, following routine primary care practices for chronic condition management. Outcomes will be compared to the intervention group over 6 months, with follow-ups at 3 and 6 months to evaluate standard diagnostic accuracy and clinical results. No additional devices or training are provided.
  Interventions: Device: Truway Portable Ultrasound Device; Device: Truway Blood Glucose Monitor; Drug: Standard Oral Hypoglycemic Agent

INTERVENTIONS:
Device: Truway Portable Ultrasound Device — Participants in the intervention group will use the Truway Portable Ultrasound Device, a FDA-regulated diagnostic tool, to perform non-invasive imaging for early detection of chronic conditions such as cardiovascular disease. The device will be used under supervised primary care protocols over a 6-month period, with training provided to care providers. Calibration and maintenance will be managed by Truway Health, Inc.
Device: Truway Blood Glucose Monitor — Participants in the intervention group will utilize the Truway Blood Glucose Monitor, an FDA-regulated device, to measure blood glucose levels for early detection and management of diabetes. The device will be employed under supervised primary care protocols over 6 months, with follow-ups at 3 and 6 months to assess accuracy and clinical outcomes. Training and support will be provided by Truway Health, Inc.
Drug: Standard Oral Hypoglycemic Agent — Participants in the intervention group with diagnosed prediabetes or Type 2 Diabetes Mellitus may receive a standard oral hypoglycemic agent (e.g., metformin) as prescribed by their primary care provider, in conjunction with the Truway diagnostic devices. The drug will be administered according to FDA-approved guidelines over the 6-month study period, with dosages adjusted based on blood glucose monitoring results obtained from the Truway Blood Glucose Monitor. Follow-ups at 3 and 6 months will assess glycemic control and safety.

SUMMARY:
This study evaluates the effectiveness of Truway Health-sourced portable diagnostic devices, including ultrasound and blood glucose monitors, in early detection of chronic conditions in outpatient primary care settings. Conducted as a prospective interventional trial, 200 participants will be assigned to use these devices versus standard care over a 6-month period. The primary outcome is improved diagnostic accuracy and patient outcomes. The study, led by Truway Health, Inc., aims to enhance accessible healthcare solutions starting at a New York site, with potential expansion to Miami.

DETAILED DESCRIPTION:
This prospective interventional study, titled "Evaluation of Truway Health-Sourced Portable Diagnostic Devices for Early Detection of Chronic Conditions in Outpatient Primary Care Settings," is designed to assess the efficacy and usability of Truway Health, Inc.'s portable diagnostic tools-specifically ultrasound and blood glucose monitoring devices-in improving early detection and management of chronic conditions such as diabetes and cardiovascular disease. Conducted by Truway Health, Inc. (www.truwayhealth.com) (www.truwayhealth.com), a leader in e-commerce medical supply distribution, the study leverages the company's expertise to address gaps in affordable, point-of-care diagnostics.The study will enroll 200 participants from a single initial site, the Truway Health Clinical Research Center in New York, NY, with plans to expand to a second site in Miami, FL, pending initial results and enrollment success. Participants, aged 18-75 with risk factors for chronic conditions (e.g., obesity, family history), will be randomly assigned to one of two groups: an intervention group using Truway-sourced devices under supervised primary care protocols, or a control group receiving standard care without these tools. The intervention period will span 6 months, with follow-up assessments at 3 and 6 months to evaluate diagnostic accuracy, patient adherence, and clinical outcomes (e.g., HbA1c levels, early detection rates).The primary objective is to determine whether Truway's portable devices enhance early detection rates compared to standard care, with secondary endpoints including cost-effectiveness, patient satisfaction, and healthcare provider feedback. Data will be collected via electronic health records and patient surveys, analyzed using statistical methods to assess significance (p<0.05). The study adheres to FDAAA 801 requirements, with results intended for public posting on ClinicalTrials.gov upon completion.Led by Principal Investigator Gavin Solomon, MD, President & CEO of Truway Health, Inc., the trial is sponsored by the company with no current U.S. Government funding. Ethical approval from an Institutional Review Board (IRB) is pending, with recruitment targeted to begin February 1, 2026. Challenges include ensuring device calibration across sites and compliance with regulatory reporting timelines. This initiative reflects Truway Health's commitment to innovative healthcare solutions, with findings potentially informing future device distribution and clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 75 years, inclusive

Ability to understand the study procedures and provide written informed consent

Diagnosis of the target condition according to established clinical or diagnostic criteria

Stable treatment regimen (pharmacologic or non-pharmacologic) for at least 4 weeks prior to screening

Willingness and ability to comply with all study visits, procedures, and follow-up assessments -

Exclusion Criteria:

Pregnancy or breastfeeding at the time of enrollment

Known hypersensitivity to any components of the investigational intervention

Uncontrolled or unstable comorbid conditions (for example, cardiovascular, hepatic, renal, or psychiatric disorders)

Participation in another interventional clinical trial within the past 3 months

Cognitive impairment or language barrier that would preclude valid informed consent or reliable reporting

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Early Detection of Chronic Conditions | 6 months
  The percentage of participants with early detection of chronic conditions (e.g., Type 2 Diabetes Mellitus, Cardiovascular Disease) using Truway Health-sourced portable diagnostic devices (ultrasound and blood glucose monitor) compared to standard care. Early detection is defined as identification of abnormalities (e.g., elevated HbA1c ≥5.7%, abnormal ultrasound findings) prior to clinical symptom onset.
Improvement in Glycemic Control | 6 months
  The change in HbA1c levels among participants with prediabetes or Type 2 Diabetes Mellitus in the intervention group using the Truway Blood Glucose Monitor and standard oral hypoglycemic agent, compared to the control group receiving standard care.

SECONDARY OUTCOMES:
Patient Satisfaction with Diagnostic Tools | 6 months
  The level of participant satisfaction with the use of Truway Health-sourced portable diagnostic devices (ultrasound and blood glucose monitor), measured using a validated satisfaction survey (e.g., Likert scale 1-5) compared to satisfaction with standard care.

CONTACTS AND LOCATIONS:
Locations (1):
- Truway Health, Inc., New York, New York, United States